CLINICAL TRIAL: NCT07349628
Title: Preoperative Botulinum Toxin A Enables Fascial Closure and Reduces Morbidity in Complex Incisional Hernias: Results From the Prospective
Brief Title: Botulinum Toxin A Facilitates Fascial Closure in Complex Incisional Hernias
Acronym: BRIDGE-HERNIA
Status: Completed | Type: Observational
Sponsor: Azienda Sanitaria Locale Napoli 2 Nord (Other)
Responsible Party: Principal Investigator, Francesco Pizza, Principal Investigator,, Azienda Sanitaria Locale Napoli 2 Nord
Other Study IDs: 18992026
Record Dates: First submitted 2026-01-06; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Incisional Hernia
Keywords: Complex incisional hernia; Ventral hernia repair; Abdominal wall reconstruction; Botulinum toxin injection; Prehabilitation
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 32 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with complex midline incisional hernia: his cohort includes adult patients with complex midline incisional hernias undergoing elective surgical repair within a standardized clinical pathway that incorporates preoperative botulinum toxin A administration. Participants are prospectively followed to collect clinical, radiological, surgical, and postoperative outcome data as part of routine clinical care.

SUMMARY:
Brief Study Description

This prospective observational study evaluates the use of preoperative botulinum toxin A as part of a structured clinical pathway for patients undergoing elective repair of complex midline incisional hernias. Botulinum toxin A is administered before surgery to temporarily relax the abdominal wall muscles, with the aim of improving abdominal wall flexibility and facilitating closure of the hernia without the need for more extensive surgical techniques. The study collects clinical, radiological, and postoperative outcome data to assess surgical feasibility, complications, and early recurrence. The overall goal is to better understand how preoperative muscle relaxation may support safer and more effective abdominal wall reconstruction.

DETAILED DESCRIPTION:
Detailed Description

This prospective observational study investigates a preoperative strategy designed to improve surgical outcomes in patients with complex midline incisional hernias. These hernias often involve large abdominal wall defects and significant muscle retraction, which can make surgical repair difficult and increase the risk of complications. To address these challenges, the study evaluates the use of botulinum toxin A administered before surgery as part of a standardized clinical pathway known as the BRIDGE-HERNIA protocol.

Botulinum toxin A is injected into the lateral abdominal wall muscles several weeks before the planned operation. Its temporary muscle-relaxing effect increases the flexibility of the abdominal wall, which may allow surgeons to close the hernia defect more easily and avoid more invasive surgical techniques. All patients undergo detailed preoperative assessment, including imaging studies, to evaluate abdominal wall anatomy and to plan the surgical approach. After botulinum toxin administration, imaging is repeated to assess changes in muscle length and hernia dimensions.

The study prospectively collects clinical, radiological, surgical, and postoperative data. Primary outcomes include the feasibility of achieving direct fascial closure without advanced component separation techniques. Secondary outcomes include postoperative complications, length of hospital stay, early hernia recurrence, and patient-reported quality of life. Because the study is observational, all treatments are delivered according to routine clinical practice, and no additional experimental interventions are assigned by the study protocol.

The results of this study aim to improve understanding of how preoperative muscle relaxation can support safer and less invasive surgical repair of complex incisional hernias, and to provide evidence that may help optimize surgical planning and patient selection in abdominal wall reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Diagnosis of complex midline incisional hernia
* Planned elective surgical repair of the incisional hernia
* Preoperative management including botulinum toxin A administration as part of routine clinical care
* Ability to undergo contrast-enhanced computed tomography imaging
* Ability to provide written informed consent

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Emergency hernia repair
  * Lateral or non-midline incisional hernia
  * Presence of true loss of domain requiring alternative surgical strategies
  * Previous allergic reaction or contraindication to botulinum toxin A
  * Neuromuscular disorders contraindicating botulinum toxin administration
  * Pregnancy or breastfeeding
  * Inability to comply with planned follow-up schedule
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Rate of fascial closure without transversus abdominis release | During surgery (index procedure)
  The proportion of patients in whom midline fascial closure is achieved using the Rives-Stoppa technique without the need for transversus abdominis release during elective repair of complex midline incisional hernias following preoperative botulinum toxin A administration.

SECONDARY OUTCOMES:
Radiological changes in abdominal wall morphology | Baseline and 5 weeks after botulinum toxin A injection
  Changes in transverse hernia defect width and lateral abdominal wall muscle elongation assessed by computed tomography before and after preoperative botulinum toxin A administration.
Postoperative complications | Up to 30 days after surgery
  Incidence of postoperative complications, including surgical site occurrences.
Length of hospital stay | Immediately after surgery
  Duration of postoperative hospital stay measured in days following elective hernia repair.
Early hernia recurrence | Up to 12 months after surgery
  Occurrence of clinically or radiologically confirmed hernia recurrence during postoperative follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Aslnapoli2Nord, Naples, Naples, Italy

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. This study is a single-center prospective observational cohort with a limited sample size, and the collected clinical and imaging data may contain potentially identifiable information. No formal data-sharing plan was included in the original study protocol, and no approval for external data sharing was obtained from the local ethics committee. Aggregate data are reported in publications, and additional information may be considered upon reasonable request and subject to institutional and ethical approval.